CLINICAL TRIAL: NCT04515797
Title: QUICKly Eradicate Hepatitis C in Patients Undergoing REnal Transplant With 4 Weeks of Glecaprevir/Pibrentasvir
Acronym: QUICK-CURE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to meet enrollment goal prior to drug expiration
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nahel Elias, M.D., Surgical Director, Kidney Transplant, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002523
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Kidney Failure; Hepatitis C; Kidney Disease, Chronic
Keywords: Kidney Transplant; Kidney Failure; HCV; Hepatitis C
MeSH Terms: conditions — Renal Insufficiency; Hepatitis C; Renal Insufficiency, Chronic | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with Direct Acting Antiviral for HCV (Experimental): 4 week treatment period with glecaprevir and pibrentasvir (G/P) within 24 hours of transplant
  Interventions: Drug: Glecaprevir and Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir and Pibrentasvir — 4 weeks of treatment starting within 24 hrs of kidney transplant
  Other Names: Direct Acting Antiviral HCV Treatment; Mavyret

SUMMARY:
This is a single center study characterizing the experience of administration of 4 weeks of pan-genotypic DAA therapy in kidney transplantation to prevent the transmission of hepatitis C virus infection from an HCV-positive donor kidney to an HCV-negative recipient.

DETAILED DESCRIPTION:
The goal of this study is to determine if the administration of glecaprevir and pibrentasvir (G/P) for 4 weeks beginning in the immediate peri-transplant period prevents establishment of HCV infection in HCV negative recipients receiving transplanted kidneys from HCV RNA positive donors.

ELIGIBILITY:
Inclusion Criteria (Recipient)

1. Met MGH Transplant Center criteria and already listed for kidney transplant with stage 5 CKD / ESRD (eGFR <15 ml/min/1.73m2 or on renal replacement therapy)
2. Must agree to birth control. Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy and at least one barrier method
3. No evidence of clinically significant liver disease at the time of transplant readiness as determined by the clinical team
4. Able to sign informed consent

Inclusion Criteria (Deceased Donor)

1. Detectable HCV NAT test
2. KDPI score is less than ≤ 0.850
3. Traditional Donor Selection Criteria Met - acceptable for transplantation per usual evaluation

Exclusion Criteria (Recipient)

1. Pregnant or nursing (lactating) women
2. HBV positivity (Ag or DNA)
3. Any contra-indication to kidney transplantation per MGH transplant center protocol
4. Any signs or symptoms of clinically significant chronic liver disease per transplant center physician
5. Inability to discontinue any medication with a known drug-drug interaction as listed in the G/P package insert

Exclusion Criteria (Deceased Donor)

1. Confirmed HIV
2. Confirmed HBV positive (surface antigen or HBV DNA positive)
3. Any standard contra-indication to donation noted in donor (significant malignancy, unusual infection, kidney anatomical damage or significant pathology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nahel Elias, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 HCV negative subjects were agreed to receive kidney transplant from HCV RNA-positive donors, resulting in 2 subjects enrolled (transplanting with an HCV RNA positive kidney). Recruitment began in May 2021 and ended in August 2023 when enrollment was closed prior to study completion.
Groups:
- Treatment With Direct Acting Antiviral for HCV: 4 week treatment period with glecaprevir and pibrentasvir (G/P) initiated within 24 hours of transplant
  Glecaprevir and Pibrentasvir: 4 weeks of treatment starting within 24 hrs of kidney transplant
Period: Overall Study
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects receiving HCV RNA positive kidney transplant and initiating treatment with DAA
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Adults receiving kidney transplant from HCV RNA positive donor [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable Blood HCV RNA Level
Description: Negative HCV RNA by blood testing at 12 weeks after the last dose of G/P
Time Frame: 12 weeks post last dose of treatment with G/P
Population: Subjects receiving at least 1 dose of G/P after receipt of donor HCV RNA positive kidney transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Adverse Events
Description: Serious and non-serious adverse events attributed to study drug and/or HCV-viremia
Time Frame: 1 Year Study Period
Population: Subjects receiving HCV RNA positive kidney transplant and initiating treatment with DAA experience protocol related adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: HCV RNA Viral Load
Description: Assessment of HCV RNA viral load at on-treatment visits, measured at both week 2 and week 4 on treatment. The viral loads measured at Week 2 and 4 are averaged together and reported in copies per mL
Time Frame: Measured at Week 2 and Week 4 of Treatment;
Population: Subjects receiving HCV RNA positive kidney transplant and initiating treatment with DAA with a negative HCV viral load at the 2 week and 4 week treatment mark of the full 4 week treatment period. For both participants, the measured HCV RNA was 0 copies/mL (no copies present in the sample/undetectable HCV RNA).
Measure: Mean (Full Range); unit: copies per mL
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 2
copies per mL | 0 [0 to 0]

4. Secondary Outcome: Allograft Function
Description: Post-transplant allograft function measured by mean eGFR over study period
Time Frame: 1 Year Study Period
Population: Data not collected
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 0

5. Secondary Outcome: Rate of Death, Graft Failure, Acute Allograft Rejection, Delayed Graft Function, ALT Elevation
Description: The rate of clinical safety outcomes: death, graft failure, acute allograft rejection, delayed graft functions, ALT elevations > 5x ULN related to study treatment with glecaprevir/Pibrentasvir
Time Frame: 1 Year Study Period
Population: Reportable outcome events in patients who 4 weeks of study treatment with glecaprevir/pibrentasvir
Measure: Mean (Full Range); unit: reported outcome events
Arm/Group | Treatment With Direct Acting Antiviral for HCV
Number analyzed (Participants) | 2
reported outcome events | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were captured beginning at DAA administration (Day 1) until 1-year post kidney transplant with HCV RNA-positive organ.
Description: For this protocol, Adverse events were defined as any untoward medical occurrence associated with administration of the DAA and/or receipt of an HCV RNA-positive kidney transplant.
Arm/Group | Treatment With Direct Acting Antiviral for HCV
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The study was closed prior to completion and prior to achieving the target of 40 participants enrolled due to the expiration of the donated investigational product (Glecaprevir / Pibrentasvir). The final study enrollment of 2 participants provides insufficient data to support analysis of all defined secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT04515797/Prot_SAP_000.pdf